CLINICAL TRIAL: NCT00340756
Title: Reproducibility of Serum Sex Steroid Measurement: A Proof of Performance Study
Brief Title: Evaluating Serum Sex Steroid Hormones
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903274; 03-C-N274; NCT00899925 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-25

CONDITIONS: Validation
Keywords: GCMS; LCMS-MS

SUMMARY:
The purpose of this study is to evaluate the reproducibility of measurements of sex hormone levels in serum samples. Researchers will collect blood from 60 healthy adults, including 20 men, 20 premenopausal women, and 20 postmenopausal women. Blood samples will be collected after study participants have fasted overnight.

DETAILED DESCRIPTION:
This evaluation of the reproducibility of serum sex steroid measurements has two components. The first is the evaluation of reproducibility of laboratory measurements of steroid sex hormones in men. This is an ancillary study to serve as a quality control (QC) measure for the ongoing DCEG Prostate Tissue Study (ORSH#: OH99-C-N025; principal investigator: Dr. Ann Hsing) so that high-quality assays can be chosen to quantify steroids in tissue. Pending satisfactory performance in serum, we will then evaluate the reproducibility of tissue hormone measurements by Gas Chromatography-Mass Spectrometry (GC-MS) or by Liquid Chromatography - Mass Spectrometry-(GC-MS) or by Liquid Chromatography- Mass Spectrometry- Mass Spectrometry (LC-MS-MS) before incorporating them into the Prostate Tissue Study. The second component of this study involves evaluation of the reproducibility of sex steroid hormone measurements in pre- and postmenopausal women. This component, although not part of the Prostate Tissue Study, is included in this summary because the laboratory, assay methods, and blood collection procedures used in the female component are identical to those in the male component and these two components will run in parallel.

The present study will evaluate the reproducibility of serum sex steroid assays using two different assay methods in different laboratories. Specifically, the study will investigate assay reproducibility at Dr. Fernand Labrie's laboratory using GC-MS and LC-MSMS and at Dr. Frank Stanczyk's laboratory using radioimmunoassay (RIA). We propose to collect overnight fasting blood from 60 healthy subjects (20 men aged 50-65, 20 premonopausal women, and 20 postmenopausal women). Once collected, the blood will be separated and aliquotted into multiple vials. Serum from each subject will be sent to Dr. Labrie, who will perform CG-MS or LC-MSMS assays, and to Dr. Stanczyk, who will perform RIA, at four different time intervals. Subject recruitment and blood collection will be performed by Westat. BBI Biotech will ship and store the specimens after they have been collected.

ELIGIBILITY:
* INCLUSION CRITERIA:

We plan to recruit healthy men aged 50-65 from Westat employees and family and friends of Westat employees.

One month later we will recruit 20 pre menopausal women (aged 20-40) and 20 post menopausal women (aged 55-75).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-08-06; Study Completion 2011-02-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States